CLINICAL TRIAL: NCT02231788
Title: A Multicenter, Prospective, Randomized, Open-label, Phase 4 Trial to Evaluate the Efficacy of Telmisartan/S-Amlodipine(Telminuvo® Tab. 40/2.5mg) on 24-hour Ambulatory BP Control Compared With Telmisartan Monotherapy in Hypertensive Patients Inadequately Controlled by Telmisartan Monotherapy
Brief Title: The Efficacy of a Combination of Telmisartan/S-Amlodipine Compared With Telmisartan Monotherapy
Acronym: TENUVA-BP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 330HT13010
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Telminuvo; Telmitrend; Hypertension; 24hr ABPM; Telmisartan; S-amlodipine
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telminuvo®Tab. 40/2.5mg (Experimental): Telminuvo®Tab.(Telmisartan/S-Amlodipine) 40/2.5mg
  Interventions: Drug: Telminuvo®Tab. 40/2.5mg
- Telmitrend®Tab. 80mg (Active Comparator): Telmitrend®Tab.(Telmisartan) 80mg
  Interventions: Drug: Telmitrend®Tab. 80mg

INTERVENTIONS:
Drug: Telminuvo®Tab. 40/2.5mg — Telminuvo®Tab. 40/2.5mg, Once daily, Per oral for 8weeks after 2~4weeks run-in period with Telmitrend®Tab. 40mg
  Other Names: Telmisartan/S-Amlodipine 40/2.5mg
  Arms: Telminuvo®Tab. 40/2.5mg
Drug: Telmitrend®Tab. 80mg — Telmitrend®Tab. 80mg, Once daily, Per oral for 8weeks after 2~4weeks run-in period with Telmitrend®Tab. 40mg
  Other Names: Telmisartan 80mg
  Arms: Telmitrend®Tab. 80mg

SUMMARY:
The Efficacy of a Fixed Dose Combination of Telmisartan/S-Amlodipine on 24-hour Ambulatory BP Control Compared with Telmisartan Monotherapy

DETAILED DESCRIPTION:
A multicenter, Prospective, Randomized, Open-label, Phase 4 Trial designed to Evaluate the Efficacy of a Fixed Dose Combination of Telmisartan/S-Amlodipine on 24-hour Ambulatory BP Control Compared with Telmisartan Monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. More than 19 years in hypertension patient
2. Hypertension is satisfied with the Clinic blood pressure that was measured at the time of randomization

   * Clinic MSSBP ≥ 140mmHg
   * Clinic MSSBP ≥ 130mmHg in diabetes mellitus or chronic kidney disease

     * Diabetes mellitus

       * Before screening, diagnosed with diabetes mellitus being treated with oral hypoglycemic agents at least 30 days OR
       * Patients who meet the following results of laboratory tests at the time of randomization. : Fasting plasma glucose ≥ 126mg/dL
     * Chronic kidney disease

       * Patients who meet the following results of laboratory tests at the time of randomization.: 15mL/min/1.73m2 ≤ estimated glomerular filtration rate ≤ 60mL/min/1.73m2
3. Patient who decided to participate and signed on an informed consent form willingly

Exclusion Criteria:

1. Clinic MSSBP ≥ 200mmHg or Clinic MSDBP ≥ 120mmHg at the time of Screening and Randomization
2. As night workers who sleep during the day and whose working hours including 00:00 to 04:00
3. Abnormal laboratory test results

   * Aspartate aminotransferase/Alanine aminotransferase > Upper normal limit X 3
   * Serum creatinine > Upper normal limit X 4
4. Secondary hypertension patient without diabetes mellitus, chronic kidney disease: coarctation of aorta, cushing's syndrome, pheochromocytoma, primary aldosteronism etc.
5. Severe heart disease(Heart failure; New York Heart Association(NYHA) class 3, 4) and recent unstable angina or myocardial infarction or valvular heart disease or arrhythmia requiring treatment within the past 3 months
6. Severe cerebrovascular disorders such as cerebral infarction, cerebral hemorrhage within 6 months
7. Patient who is planning for a renal transplantation during the trial
8. Severe or malignant retinopathy
9. Acute of chronic inflammatory status requiring treatment
10. A history of cancer within five years
11. A history of angioedema with ACE inhibitors or angiotensin-Ⅱ receptor blockers
12. Severe hypersensitivity to amlodipine or telmisartan
13. Surgical or medical conditions

    * History of major gastrointestinal surgery
    * History of active inflammatory bowel syndrome within 12 months
    * Abnormal pancreatic functions
    * Gastrointestinal/rectal bleeding
    * Urinary tract obstruction
14. Need for other antihypertensive drugs during the trial
15. Need for prohibited medication specified in the protocol
16. Administration of other Investigational Product within 30 days
17. History of drug or alcohol abuse within 6 months
18. Pregnant, breast-feeding and childbearing age who don't use adequate contraception
19. Another clinical condition in investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 24hr mean blood pressure by ambulatory blood pressure monitoring(ABPM) at week 8. | Baseline and week 8

SECONDARY OUTCOMES:
Change from baseline in the 24hr mean daytime, nighttime, morning blood pressure by ABPM at week 8. | Baseline and week 8
  Each timepoint is as following:
  * Daytime: 06:00~21:59
  * Nighttime: 22:00~05:59
  * Morning: 06:00~11:59
Change from baseline in the clinic mean blood pressure at week 8. | Baseline and week 8
24hr ABPM and Clinic BP control at week 8. | Baseline and week 8
  <24hr ABPM>
  * 24hr mean BP: 24hr mean Systolic blood pressure(SBP)<130mmHg and 24hr mean Diastolic blood pressure(DBP)<80mmHg
  * Daytime BP: Daytime mean SBP<135mmHg and Daytime mean DBP<85mmHg
  * Night time BP: Night time mean SBP<120mmHg and Night time mean DBP<70mmHg
  <Clinic BP>
  : Mean sitting systolic blood pressure(MSSBP)<140mmHg and Mean sitting diastolic blood pressure(MSDBP)<90mmHg (If Hypertension with Diabetes mellitus or Chronic kidney disease: MSSBP<130mmHg and MSDBP<80mmHg)
24hr ABPM and Clinic BP response at week 8. | Baseline and week 8
  <24hr ABPM> 24hr mean SBP and DBP reduction≥10mmHg
  <Clinic BP> MSSBP and MSDBP≥10mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, Professor, Principal Investigator — Seoul University Hospital
Locations (11):
- South Korea (11):
  - Korea University Ansan Hospital, Gyeonggi-do, Ansan-si
  - Jeju National University Hospital, Jeju City, Aran
  - Bundang Cha Hospital, Seongnam, Bundang-gu
  - Seoul University Bundang Hospital, Seongnam, Bundang-gu
  - KyungHee University Medical Center, Seoul, Dongdaemun-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Kumi cha Hospital, Gumi, Gyeongsangbuk-do
  - Seoul University Hospital, Seoul, Jongro-gu
  - National Medical Center, Seoul, Jung-gu
  - Kosin University Gospel Hospital, Busan, Seo-gu
  - Hallym University Kangnam Sacred Heart Hosipital, Seoul, Yeongdeungpo-gu

REFERENCES:
- [Derived] Kim BJ, Cho KI, Kwon HM, Choi SM, Yoon CH, Lim SW, Joo SJ, Lee NH, Lim SY, Lim SH, Kim HS. Effect of a fixed-dose combination of Telmisartan/S-amlodipine on circadian blood pressure compared with Telmisartan monotherapy: TENUVA-BP study. Clin Hypertens. 2022 Mar 1;28(1):7. doi: 10.1186/s40885-021-00184-0. PMID 35227313